CLINICAL TRIAL: NCT01289834
Title: A Migration (RSA) and Bone Density (DEXA) Study Comparing Hi-Fatigue Bone Cement and Palacos Bone Cement in Fixation of a Smooth vs. a Fine-blasted Femoral Stem. A Prospective Randomized Study on Primary Total Hip Arthroplasty.
Brief Title: A Migration and Bone Density Study Comparing Hi-Fatigue Bone Cement and Palacos Bone Cement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VEK20100112
Record Dates: First submitted 2010-09-17; First posted 2011-02-04 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Hip Arthritis
Keywords: RSA; Bone Cement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hi-Fatigue Bone Cement (Active Comparator): CPT femoral stems fixed with Hi-Fatigue Bone Cement
  Interventions: Device: Hi-Fatigue Bone Cement
- Palacos Bone Cement (Active Comparator): CPT femoral stems fixed with Palacos Bone Cement
  Interventions: Device: Palacos Bone Cement

INTERVENTIONS:
Device: Hi-Fatigue Bone Cement — Hi-Fatigue bone cement is a new development of Aap Biomaterials, GmbH & Co that has not yet been tested in the clinical setting. Hi-Fatigue has a medium to low viscosity. Laboratory tests confirm Hi-Fatigue bone cement to have properties equivalent to or better than the golden standard bone cement" Palacos. Hi-Fatigue is to be used without pre-chilling. When mixed at a room temperature of 21°C Hi-Fatigue has a low initial viscosity improving mixing and theoretically reducing the porosity of the cured cement.
  Arms: Hi-Fatigue Bone Cement
Device: Palacos Bone Cement — Palacos Bone Cement has been used for 48 years and has a good reputation as the "gold standard" among bone cements (3). It is a high-viscosity cement with rapid application that makes it advantageous for use in orthopedic joint surgery. Palacos cement was developed in order to allow hand mixing of monomers and polymers in a dish in the operating room. Air pollution with toxic monomers in the operating room was a problem that was primarily solved by exhaust ventilation, later supplemented with vacuum mixing
  Arms: Palacos Bone Cement

SUMMARY:
The purpose of this scientific study is to compare early migration of hip prostheses in respect to the bone in order to determine whether there is a clinical difference between the two investigated bone cements (which one is best suited for cementation of hip prostheses).

DETAILED DESCRIPTION:
A randomized controlled clinical trial on 50 hybrid hips age above 70 years to the described two surgical procedures will be performed at Aarhus University hospital by two orthopaedic consultants. Randomization in 10 blocks of ten patients distributed with five patients for Palacos Cement and five patients for Hi-Fatigue Cement.

* 25 CPT femoral stems fixed with Hi-Fatigue Bone Cement.
* 25 CPT femoral stems fixed with Palacos Bone Cement.

All patients will be operated by the postero-lateral approach. The post-operative treatment and training will not differ from the standard.

ELIGIBILITY:
Inclusion Criteria:

* primary hip osteoarthritis
* sufficient bone quality for total hip arthroplasty
* age 71 years and above
* no upper age limit if the patient is capable
* informed and written consent
* patient can only enter the project with one hip

Exclusion Criteria:

* planned bilateral hip surgery
* neuromuscular or vascular disease in the affected leg
* preoperatively not found suitable for a hip arthroplasty
* patients with osteoporosis based on former diagnosis or preoperative DEXA-scan
* fracture sequelae, osteonecrosis or previous extensive hip surgery
* patients who cannot refrain from taking NSAID post-operatively
* continuous medical treatment with vitamin K antagonists (Warfarin) which is known to reduce the bone mass by a factor of 5
* patients with metabolic bone disease
* patients with rheumatoid arthritis
* postmenopausal women in systemic estrogenic hormone substitution
* patients with a continuous need of systemic cortisone treatment
* non-Danish citizenship
* patients who do not comprehend the Danish language (read and speak)
* senile dementia
* alcoholism - defined as men drinking more than 21 units a week and women drinking more than 14 units a week
* drug abuse
* major psychiatric disease
* metastatic cancer disease and treatment with radiation therapy or chemotherapy
* severe systemic disease (e.g. hemi paresis and Parkinson disease)
* systemic hip and spine disease
* employee at the orthopaedic department, Aarhus University Hospital
* ongoing case regarding industrial injury insurance of the knee
* patients with poor dental status (risk of infection)

Min Age: 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2024-01 (Actual)

PRIMARY OUTCOMES:
Femoral component migration (roentgen stereo photogrammetric analysis - RSA) | 2 years
  Migration of the femoral component is measured over time and in respect to the femur bone.

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Soballe, Professor MD, Principal Investigator — Orthopaedic Center, Aarhus University Hospital
Locations (1):
- Kjeld Soballe, Orthopaedic center, University of Aarhus, Aarhus, Denmark

REFERENCES:
- [Derived] Jorgensen PB, Krag-Nielsen N, Lindgren L, Morup RMS, Kaptein B, Stilling M. Radiostereometric analysis: comparison of radiation dose and precision in digital and computed radiography. Arch Orthop Trauma Surg. 2023 Sep;143(9):5919-5926. doi: 10.1007/s00402-022-04674-0. Epub 2022 Nov 23. PMID 36422666